CLINICAL TRIAL: NCT07198243
Title: Prospective Randomized Controlled Proof-of-concept Trial to Investigate the Effects of STW 5-II on Duodenal Mucosa and Symptoms in Functional Dyspepsia
Brief Title: The Effects of STW 5-II on Duodenal Mucosa and Symptoms in Functional Dyspepsia
Acronym: DESTINY
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S70188; 2025-521141-24-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-18; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-07

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Functional dyspepsia patients taking the matching placebo for 8 weeks.
  Interventions: Drug: Placebo
- STW 5-II (Experimental): Functional dyspepsia patients taking STW 5-II, the active product for the treatment of FD.
  Interventions: Drug: STW 5-II

INTERVENTIONS:
Drug: STW 5-II — STW 5-II is an herbal medicinal product for the symptomatic treatment of functional dyspepsia with main symptoms such as epigastric pain, epigastric burning, postprandial fullness and early satiation, but often also loss of appetite, excessive belching and heartburn. STW5-II consists of six herbal extracts: bitter candy tuft, camomile flower, caraway fruit, melissa leaf, peppermint leaf, and licorice root.
  STW 5-II will be a solution for oral intake, for the treatment of FD, administered as 20 droplets in liquids, three times daily during 8 weeks. Recommended time of ingestion is just before or with meals. Patients and study staff are blinded for the intervention
  Arms: STW 5-II
Drug: Placebo — Matching placebo will be a solution for oral intake, administered as 20 droplets in liquids, three times daily during 8 weeks. Recommended time of ingestion is just before or with meals. Patients and study staff are blinded for the intervention.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to find out whether a herbal medicine called STW 5-II can help improve gut health and symptoms in adults recently diagnosed with functional dyspepsia (FD)-a condition that causes frequent stomach discomfort, especially after eating.

The main questions it aims to answer are:

Can STW 5-II reduce certain immune cells (eosinophils) in the gut lining? Can it improve symptoms like severe postprandial fullness, bloating, epigastric pain, and improve quality of life?

Researchers will compare STW 5-II to a placebo to see if it helps reduce gut inflammation and ease symptoms.

Participants will:

Take either STW 5-II or a placebo for 8 weeks Provide small samples of gut tissue (via endoscopy) Answer questions about their symptoms and daily life An optional 4-week treatment with STW 5-II will follow for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years newly to be treated with an FD/PDS diagnosis (Rome IV clinical criteria).
* Newly to be treated patients are defined as patients currently not on any ongoing treatment for FD (including OTC medication) for the last 2 weeks. Medications such as PPI or others that may affect GI function and symptom should be stopped prior the trial (min 4 weeks). See list of forbidden medication.
* Male or female using contraception or postmenopausal
* Witnessed written informed consent
* Capable to understand and comply with the study requirements

Exclusion Criteria:

Inclusion criteria:

* Patients ≥18 years newly to be treated with an FD/PDS diagnosis (Rome IV clinical criteria).
* Newly to be treated patients are defined as patients currently not on any ongoing treatment for FD (including OTC medication) for the last 2 weeks. Medications such as PPI or others that may affect GI function and symptom should be stopped prior the trial (min 4 weeks). See list of forbidden medication.
* Male or female using contraception or postmenopausal
* Witnessed written informed consent
* Capable to understand and comply with the study requirements

Exclusion criteria:

* Major active somatic or psychiatric condition that may explain dyspeptic symptoms (stable dose of single antidepressant allowed for psychiatric indication, no limitation for other indications) Predominant symptoms of gastro-esophageal reflux disease (GERD) or irritable bowel syndrome (IBS)
* Chronic ppi use. No PPI use for at least the prior 4 weeks before entering the trial- History of major abdominal surgery (except for appendectomy, cholecystectomy or splenectomy)
* History or presence of diabetes mellitus type 1 & type 2, coeliac disease or inflammatory bowel disease
* Active malignancy
* Known HIV, HBV or HCV infection
* Significant alcohol use (>10 units/weeks)
* Females pregnant or lactating
* Hypersensitivity against ingredients of STW 5-II or placebo (see annex)
* Abnormal baseline laboratory blood values

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Difference in duodenal mucosal eosinophil count between baseline and the end of the treatment (week 8) in both arms | 8 weeks
  For the primary outcome, the number of eosinophils per square mm tissue will be counted as described by Ceulemans M et al. The numbers of cells will be compared at the end of treatment between both study arms.
  The baseline values and the delta over time will also be compared between both groups. If necessary, the baseline value can be added as co-variate in the statistical analysis.

SECONDARY OUTCOMES:
The effect of STW 5-II vs. placebo therapy on clinical symptoms | 8 weeks
  The LPDS diary will be analysed using a linear mixed model on data collected up to 8 weeks, including the baseline value as a covariate and including stratum, randomised group, and time (4 weeks and 8 weeks) as fixed factors in the model. The interaction between time and group will also be included to allow for different evolutions over time for the two groups. A random intercept per patient will be included to account for interdependencies within patient. From this model, the mean difference between randomised groups at 8 weeks will be estimated and presented along with its 95% confidence interval.
The effect of STW 5-II in other immune cells | 8 weeks
  Mast cells counts will be also done and analysed as described by Ceulemans M et al. The numbers of cells will be compared at the end of treatment between both study arms. The baseline values and the delta over time will also be compared between both groups. If necessary, the baseline value can be added as co-variate in the statistical analysis.
Changes in Mucosal permeability | 8 weeks
  Changes in Mucosal permeability in transmucosal electrical resistance (TEER) and transmucosal flux of a fluorescent molecule in Ussing chambers, and tight junction proteins will be evaluated before and after treatment

OTHER OUTCOMES:
The effect of STW 5-II vs. placebo therapy on quality of life | 8 weeks
  The effect of STW 5-II vs. placebo therapy on quality of life using the Patient Assessment of Upper Gastrointestinal. Disorders-Quality Of Life instrument This is a 30 item questionnaire. Each item is scored on a 6-point Likert scale, ranging from 0 (lowest QOL) to 5 (highest QOL),
The effect of STW 5-II vs. placebo in co-morbidities (depression ) in functional dyspepsia | 8 weeks
  co-morbidity of depression using the PHQ-9 questionnaire (Patient Health Questionnaire-9) will be evaluated before vs. after treatment. The PHQ-9 (Patient Health Questionnaire-9) is a self-administered questionnaire used to screen for depression and assess its severity. It has ONE UNIT OF MEASURE, which is the total score of a 9 questions. Each of the nine questions is scored on a scale of 0-3, with 0 being "Not at all" and 3 being "Nearly every day". The total score, which can range from 0 to 27, is then interpreted to determine the level of severity of depression.
The effect of STW 5-II vs. placebo in co-morbidities (somatization) in functional dyspepsia | 8 weeks
  co-morbidity of somatization using the PHQ-15 questionnaire (Patient Health Questionnaire-15) will be evaluated before vs. after treatment. The Patient Health Questionnaire-15 (PHQ-15) assesses the severity of somatic symptoms. It has ONE UNIT OF MEASURE, which is the total score of a 15 questions. It is scored by assigning values of 0, 1, or 2 to each of the 15 items, corresponding to "not bothered at all," "bothered a little," and "bothered a lot," respectively. The total score, ranging from 0 to 30, reflects the overall severity of somatic symptoms. Higher scores indicate greater severity of somatic symptoms
The effect of STW 5-II vs. placebo in co-morbidities (anxiety) in functional dyspepsia | 8 weeks
  co-morbidity of somatization using the GAD-7 questionnaire (Generalized Anxiety Disorder 7-item scale) will be evaluated before vs. after treatment.
  The GAD-7 is a questionnaire used to screen for and assess the severity of generalized anxiety disorder. Scores range from 0 to 21, with higher scores indicating more severe anxiety. A score of 10 or more suggests a possible GAD diagnosis.
Overall treatment efficacy evaluation | 8 weeks
  The overall treatment efficacy will be evaluated before vs. after the treatment.
  AI-overzicht The Overall Treatment Effect (OTE) score, used in clinical settings, is a patient-reported outcome that measures the perceived change in symptoms or health-related quality of life (HRQoL) after a treatment. It's a 15-point scale ranging from -7 to +7, where negative scores indicate worsening symptoms, 0 indicates no change, and positive scores indicate improvement.
Overall symptom severity valuation | 8 weeks
  The overall symptom score (OSS) will be evaluated before vs. after the treatment.
  The overall symptom score (OSS) score, used in clinical settings, is a patient-reported outcome that measures the perceived change in symptoms. Symptoms are typically rated using a Likert scale, with options ranging from "no symptom" to "very severe". The scores for individual symptoms are then summed to calculate the overall symptom score

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven / UZLeuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided